CLINICAL TRIAL: NCT04321954
Title: A Phase 2 Study of Neoadjuvant Lenvatinib in Locally Advanced Invasive Thyroid Cancer
Brief Title: Lenvatinib in Locally Advanced Invasive Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Randolph, MD, Professor of Otolaryngology Head and Neck Surgery, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-524
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Differentiated Thyroid Cancer; Advanced Cancer
Keywords: Differentiated Thyroid Cancer; Advanced Cancer
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LENVATINIB (Experimental): Study procedures include screening for eligibility and study treatment, evaluations, and follow up visits
  * Lenvatinib will be administered orally daily at a predetermined dose for 2, 4, or 6 cycles, dependent on response. 1 cycle is 28 days.
  * Surgery per standard of care will follow lenvatinib treatment.
  Interventions: Drug: LENVATINIB

INTERVENTIONS:
Drug: LENVATINIB — Orally
  Other Names: Lenvima

SUMMARY:
This research is being done to evaluate the safety and efficacy of neoadjuvant lenvatinib on surgical outcomes of patients with invasive extrathyroidal differentiated thyroid cancer (DTC).

This research study involves a study drug called lenvatinib

DETAILED DESCRIPTION:
This is a multicenter, phase II, open-label study examining the effect of neoadjuvant lenvatinib being given to patients with extrathyroidal differentiated thyroid cancer (DTC) prior to surgery to remove cancerous tumors (thyroidectomy).

- The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* This research study involves a study drug called lenvatinib.
* It is anticipated that 30 people will participate in the study.

The U.S. Food and Drug Administration (FDA) has not approved lenvatinib for the specific disease of extrathyroidal differentiated thyroid cancer (DTC) but it has been approved for other uses.

Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at the time of informed consent and willing and able to provide written informed consent for the trial.
* Adult participants who are either initially diagnosed with locally advanced thyroid neoplasm or have experienced persistent or recurrent thyroid and/or cervical nodal recurrent DTC (participants with M1 disease are allowed, AJCC 8th edition stage I-IVb)), including:

  * a. Papillary thyroid carcinoma (PTC) - classical and variants

    * Follicular variant
    * Variants including but not limited to tall cell, columnar cell, cribriform-morular, solid, oxyphil, Warthin's-like, trabecular, tumor with nodular fasciitis-like stroma, Hürthle cell variant of papillary carcinoma
  * b. Follicular thyroid carcinoma (FTC)
  * c. Hürthle cell carcinoma
  * d. Poorly differentiated thyroid carcinoma
  * e. Cytologically confirmed thyroid neoplasm, Bethesda 3, 4 and 5
* Evidence of extrathyroidal extension and/or locally invasive disease and deemed at risk for R2 resection by treating team on clinical and/or fiberoptic examination and/or radiographic evaluation in the primary or recurrent setting. Evidence of "at risk for R2 resection" includes:

  * a. Vocal cord paralysis by fiberoptic examination
  * b. Extrathyroid and/or extranodal extension on CT or MRI, including tracheal and/or laryngeal cartilage invasion, esophageal involvement, and/or involvement of perithyroid muscles (e.g. strap, sternocleidomastoid, inferior constrictor muscles) or bone involvement
  * c. Extension into the mediastinum with visceral and/or vascular involvement
  * d. Involvement of the carotid artery or other major vessel by 180 degrees or more (exclusive of complete encasement)
  * e. Other factors that make the participant to be "at risk for R2 resection" may be allowed, after discussion with the study's principal investigator.
* Measurable disease by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1 and no medical contraindication to surgery.
* Adequately controlled blood pressure.

  * Blood pressure ≤150/90 with or without antihypertensive medications at screening
* Adequate end-organ function (including bone marrow, coagulation, renal, liver and cardiac) 28 days prior to the study registration as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 x institutional upper limit of normal, unless attributed to Gilberts syndrome
  * AST/ALT/Alk Phos ≤3 x institutional upper limit of normal
  * INR ≤1.5 x institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥30 mL/min per Cockcroft-Gault formulation

    * The cycle 1 day 1 labs need to re-meet eligibility criteria for treatment
* Ability to swallow pills.
* Females must not be lactating or pregnant at baseline (as documented by a negative betahuman chorionic gonadotropin [ß-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of ß-hCG. A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Note: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation.

Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after.

Exclusion Criteria:

* Diagnosis of medullary thyroid carcinoma or anaplastic (undifferentiated) thyroid carcinoma.
* Radiographically identified following findings:

  * intraluminal airway tumor
  * complete carotid encasement/infiltration
* Active hemoptysis (bright red blood ≥ 1/2 teaspoon) or other uncontrolled bleeding within 21 days prior to the study registration.
* Arterial/venous thromboembolic events in the last 12 months Treatment within 30 days prior to study registration with anticoagulant or antiplatelet therapy, apart from aspirin 81 mg daily.
* Prior radiotherapy to the neck.
* Prior treatment with lenvatinib or other VEGFR-directed therapy, including sorafenib.
* Known metastasis to central nervous system.
* Females who are pregnant or breastfeeding.
* If > 1 + proteinuria on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1g/24 h will be ineligible.
* Gastrointestinal malabsorption or any other condition that in the opinion of the investigator might affect the absorption of study drug.
* Active infection requiring treatment.
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment.
* Prolongation of corrected QT interval (QTc) to > 480 ms as demonstrated by a repeated ECG or any clinically significant ECG abnormality
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenvatinib.
* Any medical or other condition that in the opinion of the investigators would preclude participant's participation in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Overall R0/R1 resection rate | 112 Days
  Evaluate the overall R0/R1 resection rate, as defined by proportion of patients who undergo successful thyroidectomy with clear (R0) or microscopically positive surgical margins (R1).

SECONDARY OUTCOMES:
Resection rate of R0 | 112 Days
  Evaluate R0 resection rates in each of 4 pre-specified extrathyroidal anatomic target interfaces: R0=no cancer cells seen microscopically at the resection margin
Resection rate of R1 | 112 Days
  Evaluate R1 resection rates in each of 4 pre-specified extrathyroidal anatomic target interfaces: R1 cancer cells present microscopically at the resection margin (microscopic positive margin)
Change in Surgical complexity and morbidity score (SCMS) | 112 Days
  The Thyroid Neck Group Morbidity Complexity Scoring and MGH/MEE-MSK-MD Anderson (MMM) Surgical Morbidity Complexity Score (SMCS) are incorporated, specifying on scale with 5 levels of complexity and morbidity of the surgery [mild (level 0), moderate (level 1), severe (level 2), very severe (level 3), and unresectable (level 4)]. The surgical morbidity/complexity scores will be collected at enrollment, prior to surgery, and based on intraoperative findings.
  The change in SCMS will be reported as the median SCMS value. Determined by structures requiring resection, the score takes into account preoperatively radiographically defined structures judged to be requiring resection with surgical complexity of the given resection/potential for complications, and expected patient morbidity/change of function from the resection.
Primary surgery response rate | 112 Days
  Evaluate the response rate (RR) prior to primary surgery based on Response Evaluation Criteria in Solid Tumors version 1.1
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v 5.0 | Up to 18 months
  CTCAE version 5
Unresectable to resectable conversion rate | 112 Days
  The conversion rate will be summarized as frequency (%)
  -- Determined by structures requiring resection, the RGS takes into account preoperatively radiographically defined structures judged to be requiring resection with surgical complexity of the given resection/potential for complications, and expected patient morbidity/change of function from the resection.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Randolph, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary (MEEI)
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Farlow JL, McCrary HC, Sipos JA, Phay JE, Konda B, Agrawal A. Neoadjuvant dabrafenib and trametinib for functional organ preservation in recurrent BRAF V600E-mutated papillary thyroid cancer. Oral Oncol. 2023 Dec;147:106625. doi: 10.1016/j.oraloncology.2023.106625. Epub 2023 Nov 8. PMID 37948895